CLINICAL TRIAL: NCT03036800
Title: EFFECTIVENESS AND COST OF INTEGRATING A PROTOCOL WITH USE OF LIRAGLUTIDE 3.0 MG INTO AN OBESITY SERVICE: (STRIVE Study)
Brief Title: Saxenda in Obesity Services (STRIVE Study)
Acronym: STRIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0626
Record Dates: First submitted 2016-12-20; First posted 2017-01-30 (Estimated); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Weight Loss; Diabetes Mellitus
MeSH Terms: conditions — Obesity; Weight Loss; Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Prescribing Pathway (LIRA 3mg + Standard Care) (Experimental): Standard care plus targeted use of the intervention Liraglutide (LIRA) 3mg when pre-specified stopping rules for the medication apply
  Interventions: Drug: Saxenda; Other: Specialist Obesity Management Services
- Standard Care (Active Comparator): standard Tier 3 obesity specialist service care
  Interventions: Other: Specialist Obesity Management Services

INTERVENTIONS:
Drug: Saxenda — standard care plus targeted use of Liraglutide (LIRA) 3mg when pre-specified stopping rules for the medication apply. Liraglutide (Saxenda) 6 mg/mL solution for injection in pre-filled pen, administered by subcutaneous injection. Dose escalation to 3.0 mg daily (or maximum tolerated dose)
  Other Names: Liraglutide 3mg
  Arms: Targeted Prescribing Pathway (LIRA 3mg + Standard Care)
Other: Specialist Obesity Management Services — Specialist Obesity Management Services standard of care

SUMMARY:
A two year, parallel, two group, open-label, real-world randomised controlled trial (RCT) design for subjects with severe and complex obesity who are referred to a Tier 3 or equivalent specialist weight management/obesity service. Participants will be randomised to receive 1) standard care (obesity-specialist care), or 2) targeted prescribing pathway (obesity-specialist care plus targeted use of Liraglutide 3.0mg [LIRA 3mg] with pre-specified stopping rules for the medication). The aim of the study is to compare the effectiveness, budget impact, and cost-effectiveness between the two groups in a real-world setting among otherwise largely unselected patients.

DETAILED DESCRIPTION:
Summary of Trial Design A two year, parallel, two group, open-label, real-world, RCT design for patients with severe and complex obesity who are referred to a Tier 3 obesity service (including patients who are referred to a Tier 3 service as part of the bariatric surgery pathway). The total duration of participation will be 104 weeks (+/-2 weeks).

The first 52 weeks of the study (after randomisation) will determine whether using the targeted prescribing pathway in a Tier 3 setting will result in more participants attaining ≥15% weight loss compared with standard care. The second 52 weeks of the study will assess whether patients who lose ≥15% of their baseline weight by the first 52 weeks are more likely to maintain ≥15% weight loss for another 52 weeks in the targeted prescribing pathway compared with standard care. Further, budget impact, cost-effectiveness, improvement in obesity-related co-morbidities, complementary aspects of safety, effectiveness, adherence, and treatment satisfaction of both treatment groups will be assessed and compared.

Participants will be randomised in a 2:1 fashion to either the intervention (targeted prescribing pathway + standard care) or control (standard care) group (2 intervention: 1 control). The control group will receive standard care in a specialist obesity service (Tier 3 or equivalent), according to the best practice in each site and can include total or partial meal replacement strategies. The intervention group will receive the same standard care as the control group (i.e. according to the best practice in each site) plus all participants will initially receive LIRA with pre-specified stopping rules. The targeted prescribing pathway: participants who do not meet the definition of a 'early and good responder' (defined as achieving ≥5% weight loss at 16 weeks, ≥10% weight loss at 32 weeks and ≥15% weight loss at 52 weeks) will have their LIRA 3mg treatment stopped. It is important to note that all participants will be analysed in the group to which they are randomised; in particular, participants in the intervention group who stop receiving LIRA 3mg will remain in the intervention group and will continue to receive standard care for the remainder of the study as per the targeted prescribing pathway (albeit, the part of the pathway where LIRA 3mg is not prescribed; see Figure 1).

The study is intentionally designed to reflect a pragmatic "real-world" scenario and each Tier 3 provider may require a different number of visits for their programme. However, study appointments for data collection, titration reviews, application of the stopping rules of LIRA 3mg, and dispensing will be standardised for all of the five sites.

Intervention (Targeted Prescribing Pathway)

The NHS Weight Management pathway is divided into four distinct tiers:

Tier 1: health promotion Tier 2: lifestyle interventions Tier 3: specialist multidisciplinary weight management services Tier 4: bariatric surgery

Across the UK, each region has a specialist Tier 3 obesity and/or weight management service or equivalent, usually referred to as Tier 3. This includes a clinician led multidisciplinary team approach, potentially including a specialist physician, nurse, dietician, psychologist, physiotherapist, etc. From this point forwards, Tier 3 specialist weight management and/or equivalent services will be referred to as 'Tier 3' throughout the remainder of this protocol.

Participants in the intervention group will receive the same standard care as those in the control group, i.e. the best medical practice delivered by the Tier 3 service at each site. Additionally, at baseline, LIRA 3mg will be prescribed to all of the participants in the intervention group at a starting dose of 0.6mg daily. Dose escalation of Liraglutide will occur according to a pre-specified titration protocol, from 0.6mg to a maximum of 3.0mg daily. Liraglutide dose will be initiated at 0.6mg and then increased to 1.2mg in Week 2, 1.8mg in Week 3, 2.4mg in Week 4, and 3.0mg in Week 5. Participants in the intervention group will be aware that the LIRA 3mg treatment may be stopped at various time points throughout the duration of the study and that continued use of LIRA 3mg is based upon their response to the treatment in terms of them achieving pre-defined weight loss targets at 16, 32 and 52 weeks.. Specifically, participants in the intervention group will continue to be prescribed LIRA 3mg for the 104 week duration of the study, unless one of the following stopping rules applies:

1. st stopping rule: After 16 weeks (± 14 days) on the medication, only those participants who have lost ≥5% of their baseline weight will be offered further treatment with LIRA 3mg for another 16 weeks. Participants who have not met this weight loss target will have their LIRA 3mg treatment stopped but will still continue in the targeted prescribing pathway but will receive standard care only during the remainder of the study.
2. nd stopping rule: After 32 weeks (± 14 days) on the medication, only those participants who have lost ≥10% of their baseline weight and are still on treatment with LIRA 3mg will be offered another 20 weeks on LIRA 3mg. Participants who have not met this weight loss target will have their LIRA 3mg treatment stopped but will still continue in the targeted prescribing pathway but will receive standard care only during the remainder of the study.
3. rd stopping rule: After the first year of treatment (week 52; ± 14 days), only those participants who have lost ≥15% of their baseline weight and are still on treatment with LIRA 3mg will be offered another 52 weeks on LIRA 3mg. Participants who have not met this weight loss target will have their LIRA 3mg treatment stopped but will still continue in the targeted prescribing pathway but will receive standard care only during the remainder of the study.

Participants who fail to reach the pre-defined weight-loss targets to continue LIRA 3mg treatment, or who choose to stop receiving LIRA 3mg, will continue to be offered the standard care provided by the Tier 3 service. These participants will still attend the Clinical Review Visits but not the additional visits for participants who are still on LIRA 3mg (e.g. Weeks 65 & 91) because these visits will not be relevant to them; visits at Weeks 65 and 91 are intended to provide a new prescription of LIRA 3mg and to discuss adherence and any side effects;; see Appendices 2 & 3).

Participants will remain routinely in the Tier 3 service in-line with NICE guidance throughout the duration of the research study. Participants may be offered treatment options within the duration of the study, including bariatric surgery, as per NICE guidance and according to the decision of the local Tier 3 Multidisciplinary Team. Participants who have undergone bariatric surgery after randomisation will only be included in the intention to treat (ITT) analysis. This decision was made because the proportion of participants undergoing bariatric surgery is likely to be unbalanced between the treatment groups (i.e. more participants in the control group are expected to have bariatric surgery than in the targeted prescribing pathway treatment group), and thus weight loss in these individuals could unduly influence the study results. Participants who have been prescribed and start anti-obesity medication (such as Orlistat) will be ineligible for LIRA 3mg treatment.

Control (Standard Care) Participants in the control group will follow the best medical care provided by the Tier 3 service at the relevant site. This typically involves dietary advice to reduce energy intake (and may include a period of partial or total meal replacement), accompanied - if available - by a physical activity programme, both supported by behavioural change techniques with regular professional contacts. The nature of the standard care will vary between the different Tier 3 services at each site, as this is a pragmatic 'real-world' study. Clinician input will include the medical assessment of participants for severe and complicated obesity and the prescription of anti-obesity drugs (such as Orlistat) as per local Tier 3 service policy. As with the LIRA 3mg group those patients taking antihypertensive or antidepressant medication will be assessed and it will be at the clinician's discretion as to whether these medications are changed. Participants will remain routinely in the Tier 3 service in-line with NICE guidance throughout the duration of the research study. Participants may be offered treatment options within the duration of the study, including bariatric surgery, as per NICE guidance and according to the decision of the local Tier 3 Multidisciplinary Team.

ELIGIBILITY:
Inclusion Criteria:

* be aged between 18-75 years old (inclusive)
* understand written and spoken English
* be able to give in informed consent
* a body mass index ≥35 kg/m2,
* have been referred to Tier 3 weight management or equivalent service in one of the five participating sites,
* have a stable body weight (less than 5kg self-reported change during the previous 12 weeks),
* Participant must be able to meet at least one of the inclusion criteria listed below:

  1. prediabetes (defined as established diagnosis of impaired fasting glycaemia (IFG) from GP and/or established diagnosis of impaired glucose tolerance (IGT) from GP and/or HbA1C 42-47 mmol/mol (6-6.4%) without glucose lowering medications, at a blood test during the last 6 months) and/or
  2. type 2 diabetes [defined as established diagnosis of Type II diabetes from GP and/or HbA1C ≥48 mmol/mol (>6.5%) at a blood test during the last 6 months] being treated with any combination of lifestyle, metformin, sulphonylureas, thiazolidinediones (TZDs) or SGLT-2, and/or
  3. hypertension treated (defined as being on antihypertensive treatment with or without a diagnosis of hypertension from GP) or untreated (defined as Systolic Blood Pressure (SBP) ≥140 mmHg at two consecutive visits at the Tier 3 clinic), and/or
  4. obstructive sleep apnoea (on CPAP or established diagnosis of Apnoea Hypopnoea Index ≥15 at sleep studies during the last 12 months)

Exclusion Criteria:

* Diagnosis of Type 1 diabetes
* Type 2 diabetes with treatment on DPP-IV or insulin currently
* Treatment with GLP-1 receptor agonists within the last 6 months and/or have a history of GLP-1 receptor agonist intolerance.
* Treatment with anti-obesity drugs within the last 12 weeks prior to randomisation
* eGFR ≤30ml/min/1.73m2 on serum testing over the last 26 weeks
* Females referred to the clinic because of fertility problem
* Females of child bearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using or willing to use adequate contraceptive methods during the study period
* Have terminal illness
* Are not primarily responsible for their own care
* Not willing or able to give informed consent
* Any other significant disease or disorder which in the opinion of the investigator, may either put the participants at risk or may influence the result of the study or the participant's ability to participate
* Untreated or uncontrolled hypothyroidism/hyperthyroidism defined as thyroid- stimulating hormone >6 mIU/liter or <0.4 mIU/liter
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC)
* Personal history of non-familial medullary thyroid carcinoma
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Amylase levels three times higher than the upper normal range
* Obesity induced by other endocrinologic disorders (e.g. Cushing's Syndrome)
* Current or history of treatment with medications that may cause significant weight gain, within 12 weeks prior to screening, including systemic corticosteroids (except for a short course of treatment, i.e. 7-10 days), atypical antipsychotic and mood stabilizers (e.g. clozapine, olanzapine, valproic acid and its derivatives, and lithium)
* History of major depressive episode during the last 2 years
* History of initiation of antidepressants during the last 12 weeks
* Simultaneous participation in other clinical trials of investigational drugs, lifestyle or physical activity interventions.
* Previous surgical treatment for obesity (excluding liposuction if performed >1 year before trial entry)
* History of other severe psychiatric disorders
* History of known or suspected abuse of alcohol and/or narcotics
* History of major depressive episode during the last 2 years
* Simultaneous participation in other clinical trials of investigational drugs, lifestyle or physical activity interventions. Patients will only be able to take part following participation in a previous clinical trial after a wash-out period of 16 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Davies, Prof, Principal Investigator — Univesrity of Leicester
Locations (5):
- St Vincent's University Hospital, Dublin, Ireland
- United Kingdom (4):
  - NHS Greater Glasgow and Clyde West Glasgow Ambulatory Care Hospital, Glasgow
  - University Hospitals of Leicester NHS Trust, Leicester General Hospital, Leicester
  - University Hospital Aintree, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papamargaritis D, Al-Najim W, Lim JZM, Crane J, Bodicoat DH, Barber S, Lean M, McGowan B, O'Shea D, Webb DR, Wilding JPH, le Roux CW, Davies MJ. Effectiveness of integrating a pragmatic pathway for prescribing liraglutide 3.0 mg in weight management services (STRIVE study): a multicentre, open-label, parallel-group, randomized controlled trial. Lancet Reg Health Eur. 2024 Feb 9;39:100853. doi: 10.1016/j.lanepe.2024.100853. eCollection 2024 Apr. PMID 38803628
- [Derived] Papamargaritis D, Al-Najim W, Lim J, Crane J, Lean M, le Roux C, McGowan B, O'Shea D, Webb D, Wilding J, Davies MJ. Effectiveness and cost of integrating a pragmatic pathway for prescribing liraglutide 3.0 mg in obesity services (STRIVE study): study protocol of an open-label, real-world, randomised, controlled trial. BMJ Open. 2020 Feb 13;10(2):e034137. doi: 10.1136/bmjopen-2019-034137. PMID 32060156

RESULTS

PARTICIPANT FLOW:
Groups:
- Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care): Saxenda: standard care plus targeted use of Liraglutide (LIRA) 3mg when pre-specified stopping rules for the medication apply. Liraglutide (Saxenda) 6 mg/mL solution for injection in pre-filled pen, administered by subcutaneous injection. Dose escalation to 3.0 mg daily (or maximum tolerated dose).
  Plus specialist Obesity Management Services: Specialist Obesity Management Services (Tier 3) - standard of care
- Standard Care Arm: Specialist Obesity Management Services: Specialist Obesity Management Services (Tier 3) - standard of care
Period: Overall Study
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Started | 260 | 132
Week 16 | 252 | 117
Week 32 | 243 | 113
Week 52 | 237 | 110
Week 104 | 215 | 104
Completed | 201 | 93
Not Completed | 59 | 39
Not completed — Protocol Violation | 1 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0
Not completed — Tolerance | 5 | 0
Not completed — Unknown/no reason given | 50 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm | Total
Number analyzed (Participants) | 260 | 132 | 392
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 228 | 113 | 341
  >=65 years | 32 | 19 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.10 (10.81) | 51.81 (10.77) | 51.34 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 79 | 252
  Male | 87 | 53 | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 225 | 114 | 339
  Black | 13 | 11 | 24
  South Asian | 11 | 3 | 14
  Mixed/Other | 11 | 4 | 15
Weight [Mean (Standard Deviation); unit: Kg] | 129.02 (25.33) | 127.09 (21.42) | 128.37 (24.08)
BMI [Mean (Standard Deviation); unit: Kg/m2] | 46.22 (7.75) | 45.52 (7.25) | 45.99 (7.58)
Heart Rate [Mean (Standard Deviation); unit: Beats/minute] | 78.27 (11.21) | 78.37 (12.24) | 78.30 (11.55)
Waist Circumference [Mean (Standard Deviation); unit: Centimetre] | 132.44 (15.56) | 131.81 (12.95) | 132.23 (14.73)
HbA1c mmol/mol [Mean (Standard Deviation); unit: Mmol/mol] | 46.10 (13.72) | 44.71 (10.79) | 45.64 (12.82)
HbA1c % [Mean (Standard Deviation); unit: %] | 6.36 (1.27) | 6.24 (0.99) | 6.32 (1.18)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 135.77 (18.26) | 138.12 (17.79) | 136.56 (18.12)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 81.35 (10.94) | 81.99 (12.04) | 81.57 (11.31)
LDL Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 2.71 (0.84) | 2.70 (0.83) | 2.71 (0.84)
HDL Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 1.24 (0.30) | 1.25 (0.55) | 1.24 (0.40)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 4.76 (1.00) | 4.74 (0.95) | 4.75 (0.98)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 1.85 (0.94) | 1.86 (0.94) | 1.85 (0.94)
Average total MET [Mean (Standard Deviation); unit: Minutes/week] | 5246.83 (7145.63) | 5463.48 (7958.59) | 5318.24 (7412.94)
Smoking status [Count of Participants; unit: Participants]
  Never smoker | 144 | 71 | 215
  Ex-smoker | 90 | 48 | 138
  Current smoker | 25 | 13 | 38
  Missing | 1 | 0 | 1
Glycaemic Status [Count of Participants; unit: Participants]
  Normogylcaemia | 110 | 66 | 176
  Prediabetes | 42 | 20 | 62
  Diabetes remission | 9 | 3 | 12
  Diabetes | 98 | 41 | 139
  Missing | 1 | 2 | 3
Hypertension Status [Count of Participants; unit: Participants]
  Yes | 162 | 88 | 250
  No | 96 | 44 | 140
  Missing | 2 | 0 | 2
Sleep Apnoea Status [Count of Participants; unit: Participants]
  Yes | 124 | 68 | 192
  No | 113 | 54 | 167
  Missing | 23 | 10 | 33
Number of all Medications [Count of Participants; unit: Participants]
  None | 55 | 30 | 85
  One | 24 | 11 | 35
  Two | 17 | 17 | 34
  Three | 32 | 9 | 41
  Four | 24 | 7 | 31
  Five and over | 108 | 58 | 166
Number of Diabetes Medications [Count of Participants; unit: Participants]
  Does not have diabetes | 162 | 91 | 253
  None | 35 | 12 | 47
  One | 52 | 22 | 74
  Two | 9 | 6 | 15
  Three and over | 2 | 1 | 3
Number of Antihypertensive Medications [Count of Participants; unit: Participants]
  Does not have hypertension | 98 | 44 | 142
  None | 44 | 24 | 68
  One | 55 | 25 | 80
  Two | 33 | 22 | 55
  Three and over | 30 | 17 | 47
Statin Use [Count of Participants; unit: Participants]
  Yes | 70 | 31 | 101
  No | 190 | 101 | 291

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss of ≥15% From Baseline (Complete Cases)
Description: Proportion of participants with severe and complicated obesity achieving weight loss of ≥15% at 52 weeks with the use of a targeted prescribing pathway (i.e. use of LIRA 3mg according to a pre-specified protocol in combination with standard care provided in Tier 3 services) versus standard care alone in a Tier 3 service.
Time Frame: 52 weeks
Population: Complete cases population The complete cases population is defined as all randomised participants who have data available for the outcome being analysed, according to the study group to which they were randomised at baseline. Participants who had bariatric surgery during the study period were excluded from this population.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 201 | 93
Participants | 51 | 6
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥15% from baseline at 52 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.19, 95% CI 2-sided [2.09 to 12.88]

2. Primary Outcome: Weight Loss of ≥15% From Baseline (Intention to Treat)
Description: as for outcome 1
Time Frame: 52 weeks
Population: Intention to Treat population (ITT). The ITT population was all randomised participants and they were analysed according to the treatment group to which they were randomised at baseline. Missing outcome data were imputed. Participants who had bariatric surgery during the study period were included in this population.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants | 55 | 6
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.94, 95% CI 2-sided [2.45 to 14.4]

3. Primary Outcome: Weight Loss of ≥15% From Baseline (Per Protocol)
Description: as for outcome 1
Time Frame: 52 weeks
Population: Per protocol population All participants who were compliant with their randomised treatment, analysed according to the treatment group to which they were randomised. Standard care group are compliant if they complete >70% of the planned contacts in the T3 service. The intervention group are compliant if they complete >70% of the planned contacts in the T3 service, and take >70% of their prescribed LIRA 3mg. Excludes participants who had bariatric surgery during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 108 | 51
Participants | 40 | 5
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 5.04, 95% CI 2-sided [1.81 to 14.01]

4. Primary Outcome: Weight Loss of ≥15% From Baseline (Per Protocol Without Excluded Concomitant Medications)
Description: as for outcome 1
Time Frame: 52 weeks
Population: Per protocol population. All participants who were compliant with their randomised treatment, analysed according to the treatment group to which they were randomised. Standard care group are compliant if they complete >70% of the planned contacts in the T3 service. The intervention group are compliant if they complete >70% of the planned contacts in the T3 service, and take >70% of their prescribed LIRA 3mg. Excludes participants who had bariatric surgery during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 105 | 50
Participants | 40 | 5
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 5.24, 95% CI 2-sided [1.88 to 14.64]

5. Secondary Outcome: Participant Attendance at Appointments (Intention to Treat)
Description: Attended at least 70% of scheduled Tier 3 appointments by 52 weeks
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 0 | 1
  Yes | 115 | 51
  Did not attend week 52 visit | 60 | 43
  Attended week 52 visit but variable missing | 85 | 37

6. Secondary Outcome: Participant Attendance at Appointments (Intention to Treat)
Description: Attended at least 70% of scheduled Tier 3 appointments by 104 weeks
Time Frame: 104 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 0 | 0
  Yes | 92 | 46
  Did not attend week 104 visit | 117 | 66
  Attended week 104 visit but variable missing | 51 | 20

7. Secondary Outcome: Cessation of Treatment Due to Adverse Effects (Intention to Treat)
Description: Derived binary indicator showing whether participant stopped treatment with liraglutide 3mg by 52 weeks because of adverse effects (i.e., the main reason for stopping was listed as 'adverse event' or 'unable to tolerate drug'). This number does not include people who stopped treatment due to a stopping rule or reason other than an adverse effect. Only defined for participants who were currently eligible for liraglutide 3mg treatment. Participants may have stopped treatment due to adverse effects at an earlier timepoint and so the total number of 'yes' and 'no' responses is higher than the number eligible for liraglutide 3mg at the analysis time-point, i.e. if a participant stopped at week 16 due to adverse events then they would still be included in the 'yes' response.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 111 | NA — This is for Liraglutide arm only.
  Yes | 3 | NA — This is for Liraglutide arm only.
  N/A | 146 | NA — This is for Liraglutide arm only.
  Missing | 0 | NA — This is for Liraglutide arm only.

8. Secondary Outcome: Cessation of Treatment Due to Adverse Effects (Intention to Treat)
Description: Derived binary indicator showing whether participant stopped treatment with liraglutide 3mg by 104 weeks because of adverse effects (i.e., the main reason for stopping was listed as 'adverse event' or 'unable to tolerate drug'). This number does not include people who stopped treatment due to a stopping rule or reason other than an adverse effect. Only defined for participants who were currently eligible for liraglutide 3mg treatment. Participants may have stopped treatment due to adverse effects at an earlier timepoint and so the total number of 'yes' and 'no' responses is higher than the number eligible for liraglutide 3mg at the analysis time-point, i.e. if a participant stopped at week 16 due to adverse events then they would still be included in the 'yes' response.
Time Frame: 104 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 53 | NA — This is for Liraglutide arm only.
  Yes | 2 | NA — This is for Liraglutide arm only.
  N/A | 205 | NA — This is for Liraglutide arm only.
  Missing | 0 | NA — This is for Liraglutide arm only.

9. Secondary Outcome: Participant Compliance With Treatment (Intention to Treat)
Description: Derived binary indicator showing whether participant was compliant with liraglutide 3mg treatment up to 52 weeks. This was defined using the questionnaire answers as detailed in Appendix 7 of the SAP, and so includes all participants (i.e., not only those who attended the visit) up to the point when they stopped treatment or withdrew from the study.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 23 | NA — This is for Liraglutide arm only.
  Yes | 233 | NA — This is for Liraglutide arm only.
  Missing | 4 | NA — This is for Liraglutide arm only.

10. Secondary Outcome: Participant Compliance With Treatment (Intention to Treat)
Description: Derived binary indicator showing whether participant was compliant with liraglutide 3mg treatment up to 104 weeks. This was defined using the questionnaire answers as detailed in Appendix 7 of the SAP, and so includes all participants (i.e., not only those who attended the visit) up to the point when they stopped treatment or withdrew from the study.
Time Frame: 104 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 27 | NA — This is for Liraglutide arm only.
  Yes | 229 | NA — This is for Liraglutide arm only.
  Missing | 4 | NA — This is for Liraglutide arm only.

11. Secondary Outcome: Patient Stopping of Treatment (Intention to Treat)
Description: Derived binary indicator showing whether participant had stopped treatment with liraglutide 3mg at 16 weeks (due to stopping rules or other reason, such as an adverse event despite passing the stopping rule). Only defined for participants who were on liraglutide 3mg treatment at the previous time-point.
Time Frame: 16 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 181 | NA — For Liraglutide arm only.
  Yes | 79 | NA — For Liraglutide arm only.
  Missing | 0 | NA — For Liraglutide arm only.

12. Secondary Outcome: Patient Stopping of Treatment (Intention to Treat)
Description: Derived binary indicator showing whether participant had stopped treatment with liraglutide 3mg at 32 weeks (due to stopping rules or other reason, such as an adverse event despite passing the stopping rule). Only defined for participants who were on liraglutide 3mg treatment at the previous time-point.
Time Frame: 32 weeks
Population: Intention to Treat population (ITT). The ITT population was all randomised participants and they were analysed according to the treatment group to which they were randomised at baseline. Missing outcome data were imputed. Participants who had bariatric surgery during the study period were included in this population. Only includes participants who were on liraglutide 3mg treatment at the previous time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 181 | 132
Participants
  No | 110 | NA — For Liraglutide arm only.
  Yes | 71 | NA — For Liraglutide arm only.
  Missing | 0 | NA — For Liraglutide arm only.

13. Secondary Outcome: Patient Stopping of Treatment (Intention to Treat)
Description: Derived binary indicator showing whether participant had stopped treatment with liraglutide 3mg at 52 weeks (due to stopping rules or other reason, such as an adverse event despite passing the stopping rule). Only defined for participants who were on liraglutide 3mg treatment at the previous time-point.
Time Frame: 52 weeks
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 110 | 132
Participants
  No | 53 | NA — For Liraglutide arm only.
  Yes | 57 | NA — For Liraglutide arm only.
  Missing | 0 | NA — For Liraglutide arm only.

14. Secondary Outcome: Completion of Tier 3 Despite Liraglutide Cessation by 16 Weeks (Intention to Treat)
Description: Derived binary indicator showing whether participant completed 52 weeks of the Tier 3 service programme despite stopping liraglutide 3mg at 16 weeks (due to stopping rules or other reason). Only defined for participants who stopped liraglutide 3mg treatment at 16 weeks.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 60 | NA — For Liraglutide arm only.
  Yes | 19 | NA — For Liraglutide arm only.
  N/A (still using Liraglutide 3mg at 16 weeks) | 181 | NA — For Liraglutide arm only.
  Missing | 0 | NA — For Liraglutide arm only.

15. Secondary Outcome: Completion of Tier 3 Despite Liraglutide Cessation by 32 Weeks (Intention to Treat)
Description: Derived binary indicator showing whether participant completed 52 weeks of the Tier 3 service programme despite stopping liraglutide 3mg at 32 weeks (due to stopping rules or other reason). Only defined for participants who stopped liraglutide 3mg treatment at 32 weeks.
Time Frame: 52 weeks
Population: Intention to Treat population (ITT). The ITT population was all randomised participants and they were analysed according to the treatment group to which they were randomised at baseline. Missing outcome data were imputed. Participants who had bariatric surgery during the study period were included in this population. Only includes participants who stopped liraglutide 3mg treatment at 32 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 181 | 132
Participants
  No | 49 | NA — For Liraglutide arm only.
  Yes | 22 | NA — For Liraglutide arm only.
  N/A (still using Liraglutide 3mg at 32 weeks) | 110 | NA — For Liraglutide arm only.
  Missing | 0 | NA — For Liraglutide arm only.

16. Secondary Outcome: Started on Anti-obesity Drugs at 52 Weeks (Intention to Treat)
Description: Derived binary indicator showing whether participant started on anti-obesity drugs other than liraglutide (defined as a concomitant medication listing of Orlistat) at 52 weeks.
Time Frame: 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 203 | 92
  Yes | 3 | 1
  Missing | 54 | 39

17. Secondary Outcome: Started on Anti-obesity Drugs at 104 Weeks (Intention to Treat)
Description: Derived binary indicator showing whether participant started on anti-obesity drugs other than liraglutide (defined as a concomitant medication listing of Orlistat) at 104 weeks.
Time Frame: 104 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 144 | 64
  Yes | 3 | 2
  Missing | 113 | 66

18. Secondary Outcome: Referral to Other Obesity Interventions (Intention to Treat)
Description: Number of participants referred to Tier 4 for bariatric surgery over the 104 weeks study period
Time Frame: 104 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 125 | 64
  Yes | 25 | 5
  Missing | 110 | 63

19. Secondary Outcome: Referral to Other Obesity Interventions by Site (Intention to Treat)
Description: Referrals for bariatric surgery by 104 weeks, stratified by study site.
Time Frame: 104 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  Dublin | 3 | 3
  Glasgow | 0 | 0
  Leicester | 10 | 0
  Liverpool | 2 | 1
  London | 10 | 1
  Not referred / missing | 235 | 127

20. Secondary Outcome: Bariatric Surgery Completion (Intention to Treat)
Description: Number of participants who underwent bariatric surgery by 104 weeks.
Time Frame: 104 weeks
Population: Intention to Treat population (ITT). The ITT population was all randomised participants and they were analysed according to the treatment group to which they were randomised at baseline. Missing outcome data were imputed.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 260 | 132
Participants
  No | 142 | 64
  Yes | 6 | 4
  Missing | 112 | 64

21. Secondary Outcome: Weight Loss of ≥5% From Baseline (Complete Cases)
Description: Proportion of participants reaching weight loss of ≥5% from baseline, at 16 weeks.
Time Frame: 16 weeks
Population: Complete cases. The complete cases population is defined as all randomised participants who have data available for the outcome being analysed, according to the study group to which they were randomised at baseline. Participants who had bariatric surgery during the study period were excluded from this population.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 237 | 86
Participants | 186 | 34
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥5% from baseline at 16 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.12, 95% CI 2-sided [5.26 to 19.48]

22. Secondary Outcome: Weight Loss of ≥5% From Baseline (Complete Cases)
Description: Proportion of participants reaching weight loss of ≥5% from baseline, at 32 weeks.
Time Frame: 32 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 208 | 79
Participants | 158 | 34
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥5% from baseline at 32 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.17, 95% CI 2-sided [2.86 to 9.36]

23. Secondary Outcome: Weight Loss of ≥5% From Baseline (Complete Cases)
Description: Proportion of participants reaching weight loss of ≥5% from baseline, at 52 weeks.
Time Frame: 52 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 201 | 93
Participants | 127 | 29
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥5% from baseline at 52 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.16, 95% CI 2-sided [2.39 to 7.22]

24. Secondary Outcome: Weight Loss of ≥5% From Baseline (Complete Cases)
Description: Proportion of participants reaching weight loss of ≥5% from baseline, at 104 weeks.
Time Frame: 104 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 132 | 61
Participants | 62 | 17
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥5% from baseline at 104 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p = 0.010, Regression, Logistic; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.23 to 4.84]

25. Secondary Outcome: Weight Loss of ≥10% From Baseline (Complete Cases)
Description: Proportion of participants reaching weight loss of ≥10% from baseline, at 16 weeks.
Time Frame: 16 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 237 | 86
Participants | 60 | 9
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥10% from baseline at 16 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.14, 95% CI 2-sided [2.14 to 12.39]

26. Secondary Outcome: Weight Loss of ≥10% From Baseline (Complete Cases)
Description: Proportion of participants reaching weight loss of ≥10% from baseline, at 32 weeks.
Time Frame: 32 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 208 | 79
Participants | 110 | 14
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥10% from baseline at 32 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.53, 95% CI 2-sided [3.32 to 12.86]

27. Secondary Outcome: Weight Loss of ≥10% From Baseline (Complete Cases)
Description: Proportion of participants reaching weight loss of ≥10% from baseline, at 52 weeks.
Time Frame: 52 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 201 | 93
Participants | 90 | 9
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥10% from baseline at 52 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.08, 95% CI 2-sided [3.80 to 17.16]

28. Secondary Outcome: Weight Loss of ≥10% From Baseline (Complete Cases)
Description: Proportion of participants reaching weight loss of ≥10% from baseline, at 104 weeks.
Time Frame: 104 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 132 | 61
Participants | 32 | 8
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥10% from baseline at 104 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p = 0.065, Regression, Logistic; Odds Ratio (OR) = 2.28, 95% CI 2-sided [0.95 to 5.47]

29. Secondary Outcome: Weight Loss of ≥15% From Baseline (Complete Cases)
Description: Proportion of participants reaching weight loss of ≥15% from baseline at 16 weeks.
Time Frame: 16 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 237 | 86
Participants | 10 | 2
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥15% from baseline at 16 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p = 0.206, Regression, Logistic; Odds Ratio (OR) = 2.84, 95% CI 2-sided [0.56 to 14.34]

30. Secondary Outcome: Weight Loss of ≥15% From Baseline (Complete Cases)
Description: Proportion of participants reaching weight loss of ≥15% from baseline at 32 weeks.
Time Frame: 32 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 208 | 79
Participants | 32 | 5
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥32% from baseline at 16 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p = 0.023, Regression, Logistic; Odds Ratio (OR) = 3.23, 95% CI 2-sided [1.17 to 8.90]

31. Secondary Outcome: Weight Loss of ≥15% From Baseline (Complete Cases)
Description: Proportion of participants reaching weight loss of ≥15% from baseline at 104 weeks.
Time Frame: 104 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 132 | 61
Participants | 15 | 2
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥15% from baseline at 104 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p = 0.070, Regression, Logistic; Odds Ratio (OR) = 4.11, 95% CI 2-sided [0.89 to 18.93]

32. Secondary Outcome: Maintenance of ≥15% Weight Loss Until 104 Weeks (Complete Cases)
Description: Proportion of participants maintaining weight loss of ≥15% among those who lost ≥15% at 52 weeks
Time Frame: 104 weeks
Population: Complete cases population The complete cases population is defined as all randomised participants who have data available for the outcome being analysed, according to the study group to which they were randomised at baseline. Participants who had bariatric surgery during the study period will be excluded from this population.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 41 | 5
Participants | 12 | 2
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 31, analysis 1]; Test type: Superiority; p = 0.601, Regression, Logistic; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.08 to 4.24]

33. Secondary Outcome: Absolute Weight Change (Complete Cases)
Description: Absolute change in weight (kg) from baseline
Time Frame: 16 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 237 | 86
kg | -9.61 (5.38) | -5.54 (5.87)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of absolute weight change (kg) from baseline at 16 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -4.63, 95% CI 2-sided [-5.85 to -3.4]

34. Secondary Outcome: Absolute Weight Change (Complete Cases)
Description: Absolute change in weight (kg) from baseline
Time Frame: 32 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 208 | 79
kg | -11.27 (7.70) | -5.70 (7.16)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of absolute weight change (kg) from baseline at 32 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -5.89, 95% CI 2-sided [-7.76 to -4.02]

35. Secondary Outcome: Absolute Weight Change (Complete Cases)
Description: Absolute change in weight (kg) from baseline
Time Frame: 52 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 201 | 93
kg | -10.15 (9.45) | -3.21 (8.66)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of absolute weight change (kg) from baseline at 52 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -6.87, 95% CI 2-sided [-9.03 to -4.71]

36. Secondary Outcome: Absolute Weight Change (Complete Cases)
Description: Absolute change in weight (kg) from baseline
Time Frame: 104 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 132 | 61
kg | -6.51 (9.28) | -1.27 (10.30)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of absolute weight change (kg) from baseline at 104 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -5.44, 95% CI 2-sided [-8.34 to -2.53]

37. Secondary Outcome: Percentage Weight Change (Complete Cases)
Description: Percentage change in weight from baseline
Time Frame: 16 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 237 | 86
percentage | -7.63 (4.02) | -4.39 (4.45)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of relative weight change (%) from baseline at 16 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -3.72, 95% CI 2-sided [-4.63 to -2.80]

38. Secondary Outcome: Percentage Weight Change (Complete Cases)
Description: Percentage change in weight from baseline
Time Frame: 32 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 208 | 79
percentage | -9.00 (5.82) | -4.58 (5.74)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of relative weight change (%) from baseline at 32 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -4.70, 95% CI 2-sided [-6.14 to -3.25]

39. Secondary Outcome: Percentage Weight Change (Complete Cases)
Description: Percentage change in weight from baseline
Time Frame: 52 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 201 | 93
percentage | -8.13 (7.21) | -2.67 (6.79)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of relative weight change (%) from baseline at 52 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -5.37, 95% CI 2-sided [-7.02 to -3.71]

40. Secondary Outcome: Percentage Weight Change (Complete Cases)
Description: Percentage change in weight from baseline
Time Frame: 104 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 132 | 61
percentage | -5.18 (7.47) | -1.21 (8.16)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of relative weight change (%) from baseline at 104 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p = 0.001, Regression, Linear; Mean Difference (Net) = -4.10, 95% CI 2-sided [-6.42 to -1.77]

41. Secondary Outcome: Absolute BMI Change (Complete Cases)
Description: Absolute change in BMI (kg/m2) from baseline
Time Frame: 52 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 180 | 80
kg/m2 | -3.84 (3.29) | -1.17 (2.84)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of absolute BMI change (kg/m2) from baseline at 52 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -2.7, 95% CI 2-sided [-3.5 to -1.91]

42. Secondary Outcome: Absolute BMI Change (Complete Cases)
Description: Absolute change in BMI (kg/m2) from baseline
Time Frame: 104 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 132 | 61
kg/m2 | -2.30 (3.29) | -0.49 (3.57)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of absolute BMI change (kg/m2) from baseline at 104 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -1.89, 95% CI 2-sided [-2.91 to -0.86]

43. Secondary Outcome: Absolute Waist Circumference Change (Complete Cases)
Description: Absolute change in waist circumference (cm) from baseline
Time Frame: 52 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Centimetres
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 137 | 58
Centimetres | -8.88 (7.89) | -5.58 (8.48)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of absolute waist circumference change (cm) from baseline at 52 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p = 0.01, Regression, Linear; Mean Difference (Net) = -3.28, 95% CI 2-sided [-5.77 to -0.80]

44. Secondary Outcome: Absolute Waist Circumference Change (Complete Cases)
Description: Absolute change in waist circumference (cm) from baseline
Time Frame: 104 weeks
Measure: Mean (Standard Deviation); unit: Centimetres
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 101 | 48
Centimetres | -6.42 (8.44) | -0.93 (12.54)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A linear regression model was fitted for the continuous outcome of absolute waist circumference change (cm) from baseline at 104 weeks. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p = 0.003, Regression, Linear; Mean Difference (Net) = -5.51, 95% CI 2-sided [-9.09 to -1.94]

45. Secondary Outcome: Kings College Obesity Staging (KCOS) Score (Complete Cases)
Description: Kings College Obesity Staging (KCOS) score; range 0 to 3. A higher value corresponds with higher complications and worse outcomes.
Time Frame: 52 weeks
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 145 | 63
Participants
  Normal health at baseline | 0 | 0
  Normal health at follow-up | 1 | 0
  At risk of disease at baseline | 6 | 5
  At risk of disease at follow-up | 23 | 12
  Established disease at baseline | 97 | 41
  Established disease at follow-up | 108 | 43
  Advanced disease at baseline | 42 | 17
  Advanced disease at follow-up | 13 | 8

46. Secondary Outcome: Kings College Obesity Staging (KCOS) Score (Complete Cases)
Description: as for outcome 45
Time Frame: 104 weeks
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 115 | 51
Participants
  Normal health at baseline | 0 | 0
  Normal health at follow-up | 2 | 0
  At risk of disease at baseline | 5 | 4
  At risk of disease at follow-up | 16 | 10
  Established disease at baseline | 84 | 37
  Established disease at follow-up | 86 | 35
  Advanced disease at baseline | 26 | 10
  Advanced disease at follow-up | 11 | 6

47. Secondary Outcome: Patient Health Questionnaire-9 (Complete Cases)
Description: Patient health questionnaire-9 (PHQ-9) score; range 0 to 27. A higher value corresponds with higher complications and worse outcomes.
Time Frame: 52 weeks
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 139 | 63
Participants
  Minimal depression at baseline | 27 | 16
  Minimal depression at follow-up | 48 | 24
  Mild depression at baseline | 33 | 15
  Mild depression at follow-up | 30 | 9
  Moderate depression at baseline | 29 | 23
  Moderate depression at follow-up | 27 | 14
  Moderately severe depression at baseline | 32 | 2
  Moderately severe depression at follow-up | 18 | 6
  Severe depression at baseline | 18 | 7
  Severe depression at follow-up | 16 | 10

48. Secondary Outcome: Patient Health Questionnaire-9 (Complete Cases)
Description: as for outcome 47
Time Frame: 104 weeks
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 102 | 50
Participants
  Minimal depression at baseline | 19 | 15
  Minimal depression at follow-up | 32 | 17
  Mild depression at baseline | 27 | 10
  Mild depression at follow-up | 26 | 16
  Moderate depression at baseline | 20 | 18
  Moderate depression at follow-up | 21 | 10
  Moderately severe depression at baseline | 23 | 3
  Moderately severe depression at follow-up | 12 | 4
  Severe depression at baseline | 13 | 4
  Severe depression at follow-up | 11 | 3

49. Secondary Outcome: Epworth Sleepiness Scale (Complete Cases)
Description: Epworth sleepiness scale, used to diagnose obstructive sleep apnoea; scale 0 to 24.
  A higher value corresponds with a worse outcome.
Time Frame: 52 weeks
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 145 | 62
Participants
  No obstructive sleep apnoea at baseline | 111 | 47
  No obstructive sleep apnoea at follow-up | 119 | 50
  Possible obstructive sleep apnoea at baseline | 34 | 15
  Possible obstructive sleep apnoea at follow-up | 26 | 12

50. Secondary Outcome: Epworth Sleepiness Scale (Complete Cases)
Description: as for outcome 49
Time Frame: 104 weeks
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 110 | 55
Participants
  No obstructive sleep apnoea at baseline | 85 | 38
  No obstructive sleep apnoea at follow-up | 90 | 44
  Possible obstructive sleep apnoea at baseline | 25 | 17
  Possible obstructive sleep apnoea at follow-up | 20 | 11

51. Secondary Outcome: Stop Bang Questionnaire (Complete Cases)
Description: Stop Bang questionnaire, used to diagnose obstructive sleep apnoea; scale 0 to 8.
  A higher value corresponds with a worse outcome.
Time Frame: 52 weeks
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 93 | 44
Participants
  No obstructive sleep apnoea at baseline | 10 | 4
  No obstructive sleep apnoea at follow-up | 18 | 10
  Possible obstructive sleep apnoea at baseline | 34 | 12
  Possible obstructive sleep apnoea at follow-up | 43 | 14
  Likely obstructive sleep apnoea at baseline | 49 | 28
  Likely obstructive sleep apnoea at follow-up | 32 | 20

52. Secondary Outcome: Stop Bang Questionnaire (Complete Cases)
Description: as for outcome 51
Time Frame: 104 weeks
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 84 | 40
Participants
  No obstructive sleep apnoea at baseline | 11 | 3
  No obstructive sleep apnoea at follow-up | 12 | 4
  Possible obstructive sleep apnoea at baseline | 26 | 13
  Possible obstructive sleep apnoea at follow-up | 38 | 13
  Likely obstructive sleep apnoea at baseline | 47 | 24
  Likely obstructive sleep apnoea at follow-up | 34 | 23

53. Secondary Outcome: Glycaemic Status (Complete Cases)
Description: Glycaemic status, as determined by plasma glucose concentration. The glycaemic status definition states that a participant cannot be categorised as 'diabetes remission' if they are currently using liraglutide 3mg, which means that the absence of diabetes remission cases at follow-up in the intervention group is partly by definition of glycaemic status.
Time Frame: 52 weeks
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 165 | 56
Participants
  Normoglycaemia at baseline | 52 | 24
  Normoglycaemia at follow-up | 67 | 24
  Prediabetes at baseline | 21 | 9
  Prediabetes at follow-up | 10 | 7
  Diabetes remission at baseline | 8 | 2
  Diabetes remission at follow-up | 0 | 2
  Diabetes at baseline | 84 | 21
  Diabetes at follow-up | 88 | 23

54. Secondary Outcome: Glycaemic Status (Complete Cases)
Description: as for outcome 53
Time Frame: 104 weeks
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 101 | 46
Participants
  Normoglycaemia at baseline | 25 | 19
  Normoglycaemia at follow-up | 31 | 15
  Prediabetes at baseline | 13 | 7
  Prediabetes at follow-up | 8 | 8
  Diabetes remission at baseline | 5 | 1
  Diabetes remission at follow-up | 0 | 1
  Diabetes at baseline | 58 | 19
  Diabetes at follow-up | 62 | 22

55. Secondary Outcome: HbA1c ≤7% for Those With Diabetes at Baseline (Complete Cases)
Description: Proportion of participants HbA1c ≤7% at 52 weeks, among those with diabetes at baseline.
Time Frame: 52 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 54 | 17
Participants
  No | 10 | 11
  Yes | 44 | 6

56. Secondary Outcome: HbA1c ≤7% for Those With Diabetes at Baseline (Complete Cases)
Description: Proportion of participants HbA1c ≤7% at 104 weeks, among those with diabetes at baseline.
Time Frame: 104 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 39 | 17
Participants
  No | 10 | 10
  Yes | 29 | 7

57. Secondary Outcome: HbA1c ≤6.5% for Those With Diabetes at Baseline (Complete Cases)
Description: Proportion of participants HbA1c ≤6.5% at 52 weeks, among those with diabetes at baseline.
Time Frame: 52 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 54 | 17
Participants
  No | 17 | 14
  Yes | 37 | 3

58. Secondary Outcome: HbA1c ≤6.5% for Those With Diabetes at Baseline (Complete Cases)
Description: Proportion of participants HbA1c ≤6.5% at 104 weeks, among those with diabetes at baseline.
Time Frame: 104 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 39 | 17
Participants
  No | 16 | 12
  Yes | 23 | 5

59. Secondary Outcome: Hypertension (Complete Cases)
Description: Proportion of participants with hypertension at 52 weeks.
Time Frame: 52 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 172 | 80
Participants
  Hypertension at baseline: No | 37 | 20
  Hypertension at baseline: Yes | 135 | 60
  Hypertension at follow-up: No | 41 | 21
  Hypertension at follow-up: Yes | 131 | 59

60. Secondary Outcome: Hypertension (Complete Cases)
Description: Proportion of participants with hypertension at 104 weeks.
Time Frame: 104 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 127 | 58
Participants
  Hypertension at baseline: No | 35 | 16
  Hypertension at baseline: Yes | 92 | 42
  Hypertension at follow-up: No | 38 | 15
  Hypertension at follow-up: Yes | 89 | 43

61. Secondary Outcome: Weight Loss of ≥5% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥5% from baseline at 16 weeks.
Time Frame: 16 weeks
Population: Responder population The Responder population is defined as all participants in the intervention group who achieved ≥15% weight loss at 52 weeks, and all participants in the standard care group. Participants were analysed according to the treatment group to which they were randomised at baseline. Participants who had bariatric surgery during the study period were excluded from this population.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 54 | 86
Participants | 54 | 34

62. Secondary Outcome: Weight Loss of ≥5% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥5% from baseline at 32 weeks.
Time Frame: 32 weeks
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 53 | 79
Participants | 53 | 34

63. Secondary Outcome: Weight Loss of ≥5% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥5% from baseline at 52 weeks.
Time Frame: 52 weeks
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 51 | 93
Participants | 51 | 29

64. Secondary Outcome: Weight Loss of ≥5% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥5% from baseline at 104 weeks.
Time Frame: 104 weeks
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 42 | 61
Participants | 33 | 17
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.53, 95% CI 2-sided [3.83 to 28.97]

65. Secondary Outcome: Weight Loss of ≥10% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥10% from baseline at 16 weeks.
Time Frame: 16 weeks
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 54 | 86
Participants | 34 | 9
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 23.1, 95% CI 2-sided [7.55 to 70.67]

66. Secondary Outcome: Weight Loss of ≥10% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥10% from baseline at 32 weeks.
Time Frame: 32 weeks
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 53 | 79
Participants | 53 | 14

67. Secondary Outcome: Weight Loss of ≥10% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥10% from baseline at 52 weeks.
Time Frame: 52 weeks
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 51 | 93
Participants | 51 | 9

68. Secondary Outcome: Weight Loss of ≥10% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥10% from baseline at 104 weeks.
Time Frame: 104 weeks
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 42 | 61
Participants | 23 | 8
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.71, 95% CI 2-sided [2.75 to 21.60]

69. Secondary Outcome: Weight Loss of ≥15% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥15% from baseline at 16 weeks.
Time Frame: 16 weeks
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 54 | 86
Participants | 8 | 2
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.032, Regression, Logistic; Odds Ratio (OR) = 6.14, 95% CI 2-sided [1.16 to 32.32]

70. Secondary Outcome: Weight Loss of ≥15% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥15% from baseline at 32 weeks.
Time Frame: 32 weeks
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 53 | 79
Participants | 24 | 5
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of weight loss of ≥15% from baseline at 32 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 11.48, 95% CI 2-sided [3.80 to 34.67]

71. Secondary Outcome: Weight Loss of ≥15% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥15% from baseline at 52 weeks.
Time Frame: 52 weeks
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 51 | 93
Participants | 51 | 6

72. Secondary Outcome: Weight Loss of ≥15% From Baseline (Responder Population)
Description: Proportion of participants reaching weight loss of ≥15% from baseline at 104 weeks.
Time Frame: 104 weeks
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 42 | 61
Participants | 12 | 2
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 31, analysis 1]; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 13.63, 95% CI 2-sided [2.47 to 75.09]

73. Secondary Outcome: Maintenance of ≥15% Weight Loss Until 104 Weeks (Responder Population)
Description: Proportion of participants who maintained weight loss of ≥15% among those who lost ≥15% at 52 weeks.
Time Frame: 104 weeks
Population: Complete cases. All individuals in both arms (intervention and control group) who have data available for the outcome being analysed (proportion of participants who maintained at 104 weeks weight loss of >=15% among those who lost >=15% weight loss at 52 weeks) according to the study group to which they were randomised. Participants who had bariatric surgery during the study period were excluded from this population.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 41 | 5
Participants | 12 | 2
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; A logistic regression with a binary outcome of maintenance of weight loss of ≥15% at 104 weeks was fitted. The main covariate was randomised arm, with the model also being adjusted for the stratification variables: site and baseline body mass index (≥45kg/m2; <45kg/m2); Test type: Superiority; p = 0.601, Regression, Logistic; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.08 to 4.24]

74. Secondary Outcome: Percentage Weight Change (Responder Population)
Description: Percentage change in weight from baseline
Time Frame: 16 weeks
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 54 | 86
percentage | -11.45 (3.62) | -4.39 (4.45)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 37, analysis 1]; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -6.55, 95% CI 2-sided [-7.81 to -5.29]

75. Secondary Outcome: Percentage Weight Change (Responder Population)
Description: Percentage change in weight from baseline
Time Frame: 32 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 53 | 79
percentage | -14.82 (3.85) | -4.58 (5.74)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 38, analysis 1]; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -9.59, 95% CI 2-sided [-11.30 to -7.88]

76. Secondary Outcome: Percentage Weight Change (Responder Population)
Description: Percentage change in weight from baseline
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 51 | 93
percentage | -17.21 (2.43) | -2.67 (6.79)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 39, analysis 1]; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -13.51, 95% CI 2-sided [-15.51 to -11.51]

77. Secondary Outcome: Percentage Weight Change (Responder Population)
Description: Percentage change in weight from baseline
Time Frame: 104 weeks
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 42 | 61
percentage | -11.01 (6.70) | -1.21 (8.16)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 40, analysis 1]; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -9.30, 95% CI 2-sided [-12.35 to -6.26]

78. Secondary Outcome: Absolute BMI Change (Responder Population)
Description: Absolute change in BMI (kg/m2) from baseline
Time Frame: 52 weeks
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 50 | 80
kg/m2 | -7.65 (1.65) | -1.17 (2.84)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 41, analysis 1]; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -6.16, 95% CI 2-sided [-7.03 to -5.28]

79. Secondary Outcome: Absolute BMI Change (Responder Population)
Description: Absolute change in BMI (kg/m2) from baseline
Time Frame: 104 weeks
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 42 | 61
kg/m2 | -4.86 (2.91) | -0.49 (3.57)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 42, analysis 1]; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = -4.22, 95% CI 2-sided [-5.56 to -2.89]

80. Secondary Outcome: Absolute Waist Circumference Change (Responder Population)
Description: Absolute change in waist circumference (cm) from baseline
Time Frame: 52 weeks
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: Centimetres
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 42 | 58
Centimetres | -15.33 (6.02) | -5.58 (8.48)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 43, analysis 1]; Test type: Superiority; p < 0.001, Regression, Linear; Median Difference (Net) = -8.80, 95% CI 2-sided [-11.96 to -5.64]

81. Secondary Outcome: Absolute Waist Circumference Change (Responder Population)
Description: Absolute change in waist circumference (cm) from baseline
Time Frame: 104 weeks
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: Centimetres
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
Number analyzed (Participants) | 34 | 48
Centimetres | -10.20 (8.42) | -0.93 (12.54)
Statistical Analysis 1: Comparison: Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) vs Standard Care Arm; [analysis description as in outcome 44, analysis 1]; Test type: Superiority; p = 0.001, Regression, Linear; Median Difference (Net) = -9.59, 95% CI 2-sided [-14.91 to -4.27]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the study (BL-Wk104) whether serious or not. Members of research team asked participants about AEs at each study visit and recorded these on AE/SAE logs and reported SAEs as per sponsor and regulatory requirements.
Arm/Group | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) | Standard Care Arm
All-Cause Mortality (participants affected / at risk) | 2/260 | 0/132
Serious Adverse Events (participants affected / at risk) | 43/260 | 16/132
Other Adverse Events (participants affected / at risk) | 238/260 | 89/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) (N=260) | Standard Care Arm (N=132)
Abdominal infection (Infections and infestations) | 1 (1) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bile duct infections and inflammations (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hernia Repair (Surgical and medical procedures) | 2 (2) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Febrile infection (General disorders) | 1 (1) | 1 (1)
Limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Transient cerebrovascular event (Nervous system disorders) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vulvovaginal disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Posterior pituitary disorder (Endocrine disorders) | 0 (0) | 1 (1)
Renal lithiasis (Renal and urinary disorders) | 1 (2) | 0 (0)
Auscultation (Investigations) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal vascular occlusion and infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Female reproductive tract disorder (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 3 (3) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nail operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Therapeutic procedure (Surgical and medical procedures) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide Arm - Targeted Prescribing Pathway (LIRA 3mg + Standard Care) (N=260) | Standard Care Arm (N=132)
Diarrhoea (Gastrointestinal disorders) | 72 (92) | 8 (8)
Ear infection (Infections and infestations) | 5 (6) | 10 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 34 (43) | 15 (16)
Headache (Nervous system disorders) | 38 (49) | 2 (2)
Asthenic conditions (General disorders) | 30 (32) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 38 (44) | 0 (0)
Flatulence (Gastrointestinal disorders) | 33 (39) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 37 (48) | 5 (6)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 93 (117) | 12 (12)
Nausea (Gastrointestinal disorders) | 109 (183) | 5 (5)
Influenza (Infections and infestations) | 14 (15) | 5 (5)
Lower respiratory tract infection (Infections and infestations) | 41 (63) | 17 (22)
Upper respiratory tract infection (Infections and infestations) | 18 (19) | 8 (8)
Urinary tract infection (Infections and infestations) | 21 (26) | 5 (8)
Viral infection (Infections and infestations) | 36 (41) | 7 (8)
Neurological symptom (Nervous system disorders) | 27 (31) | 6 (6)

LIMITATIONS AND CAVEATS:
Although the trial was not interrupted during COVID-19 we did issue an USM to the REC & MHRA during the pandemic to explain that certain aspects of the trial would not be possible, however measures were put in place to ensure participant safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT03036800/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT03036800/SAP_001.pdf